CLINICAL TRIAL: NCT03732820
Title: A Randomised, Double-blind, Placebo-controlled, Multicentre Phase III Study of Olaparib Plus Abiraterone Relative to Placebo Plus Abiraterone as First-line Therapy in Men With Metastatic Castration-resistant Prostate Cancer (PROpel Study)
Brief Title: Study on Olaparib Plus Abiraterone as First-line Therapy in Men With Metastatic Castration-resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D081SC00001; 2018-002011-10 (EudraCT Number)
Record Dates: First submitted 2018-09-28; First posted 2018-11-07 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer (mCRPC)
MeSH Terms: interventions — olaparib; Abiraterone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- olaparib plus abiraterone (Experimental): Olaparib is available as a film-coated tablet containing 100 milligrams (mg) or 150 milligrams (mg) of olaparib. Subjects will be administered olaparib orally at a dose of 300 milligrams (mg) twice daily (bid). The initial dosage of 300 milligrams (mg) twice daily will be composed of 2 x 150 milligrams (mg) tablets per dose. The 100 milligrams (mg) and 150 milligrams (mg) tablets will be used to manage dose reductions during the study.
  Abiraterone acetate with prednisone or prednisolone will be sourced locally as commercially available materials. Subjects will be administered abiraterone orally at a dose of 1000 milligrams (mg) once daily, in combination with prednisone or prednisolone 5 milligrams (mg) administered orally twice daily.
  Interventions: Drug: olaparib; Drug: abiraterone acetate
- placebo plus abiraterone (Placebo Comparator): Placebo to match olaparib is available as a film-coated tablet in 100 milligrams (mg) or 150 milligrams (mg). Subjects will be administered placebo orally at a dose of 300 milligrams (mg) twice daily (bid). The initial dosage of 300 milligrams (mg) twice daily will be composed of 2 x 150 milligrams (mg) tablets per dose. The 100 milligrams (mg) and 150 milligrams (mg) tablets will be used to manage dose reductions during the study.
  Abiraterone acetate with prednisone or prednisolone will be sourced locally as commercially available materials. Subjects will be administered abiraterone orally at a dose of 1000 milligrams (mg) once daily, in combination with prednisone or prednisolone 5 milligrams (mg) administered orally twice daily.
  Interventions: Drug: abiraterone acetate

INTERVENTIONS:
Drug: olaparib — 300 mg (2 x 150 milligrams (mg) tablets) twice daily
  Other Names: Lynparza
  Arms: olaparib plus abiraterone
Drug: abiraterone acetate — 1000 milligrams (mg) once daily
  Other Names: Zytiga

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety (including evaluating side effects) of combination of olaparib and abiraterone versus placebo and abiraterone in patients with metastatic castration-resistant prostate cancer (mCRPC) who have received no prior cytotoxic chemotherapy or new hormonal agents (NHAs) at metastatic castration-resistant prostate cancer (mCRPC) stage.

DETAILED DESCRIPTION:
PROpel is a phase III study evaluating the efficacy, safety, and tolerability of olaparib versus placebo when given in addition to abiraterone to patients with metastatic castration-resistant prostate cancer (mCRPC) who have not received prior chemotherapy or new hormonal agents (NHAs) for metastatic castration-resistant prostate cancer (mCRPC) (first-line setting).

Approximately 720 patients globally were planned to be randomized in PROpel in a 1:1 ratio to treatment with either olaparib and abiraterone or placebo and abiraterone. Enrolment had completed with a total of 796 patients randomised. Following the completion of global enrolment, the China cohort will randomise approximately 108 additional patients at sites in China, also in a 1:1 ratio.

Patients will receive oral treatment with olaparib 300 mg twice daily + abiraterone 1000 mg once daily or placebo twice daily + abiraterone 1000 mg once daily. Patients in both treatment groups will also receive either prednisone or prednisolone 5 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in the study protocol.
2. Provision of signed and dated, written informed consent form prior to any mandatory study specific procedures, sampling, and analyses.
3. For inclusion in i) the optional exploratory genetic research and ii) the optional biomarker research, patients must fulfill the following criteria:

   * Provision of informed consent for genetic research prior to collection of sample.
   * Provision of informed consent for biomarker research prior to collection of sample.

   If a patient declines to participate in the optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.
4. Patients must be ≥18 years of age (or ≥19 years of age in South Korea) at the time of signing the informed consent form. For patients enrolled in Japan who are <20 years of age, written informed consent should be obtained from the patient and from his legally acceptable representative.
5. Histologically or cytologically confirmed prostate adenocarcinoma.
6. Metastatic status defined as at least 1 documented metastatic lesion on either a bone scan or a computed tomography(CT)/ magnetic resonance imaging (MRI) scan.
7. First-line metastatic castration-resistant prostate cancer (mCRPC).
8. Ongoing androgen deprivation with gonadotropin-releasing hormone analogue or bilateral orchiectomy, with serum testosterone <50 nanograms per decilitre (ng/dL) (<2.0 nanomoles per litre (nmol/L)) within 28 days before randomisation. Patients receiving androgen deprivation therapy (ADT) at study entry should continue to do so throughout the study.
9. Candidate for abiraterone therapy with documented evidence of progressive disease.
10. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment.
11. Eastern Cooperative Oncology Group (ECOG) performance status 0-1, with no deterioration over the previous 2 weeks.
12. The participant has, in the opinion of the investigator, a life expectancy of at least 6 months.
13. Prior to randomisation, sites must confirm availability of either an archival formalin fixed, paraffin embedded (FFPE) tumour tissue sample, or a new biopsy taken during the screening window, which meets the minimum pathology and sample requirements in order to enable homologous recombination repair (HRR) status subgroup analysis of the primary endpoint radiographic progression-free survival (rPFS). If there is not written confirmation of the availability of tumour tissue prior to randomisation, the patient is not eligible for the study.
14. Male patients must use a condom during treatment and for 3 months after the last dose of olaparib+abiraterone when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential.

Exclusion Criteria:

1. Has a known additional malignancy that has had progression or has required active treatment in the last 5 years.
2. Patients with myelodysplastic syndrome (MDS)/ acute myeloid leukaemia (AML) or with features suggestive of yelodysplastic syndrome (MDS)/ acute myeloid leukaemia (AML).
3. Clinically significant cardiovascular disease Association Class II-IV heart failure or cardiac ejection fraction measurement of <50% during screening as assessed by echocardiography or multigated acquisition scan.
4. Planned or scheduled cardiac surgery or percutaneous coronary intervention procedure.
5. Prior revascularisation procedure (significant coronary, carotid, or peripheral artery stenosis).
6. Uncontrolled hypertension (systolic blood pressure (BP) ≥160 millimeters of mercury (mmHg) or diastolic blood pressure (BP) ≥95 millimeters of mercury (mmHg)).
7. History of uncontrolled pituitary or adrenal dysfunction.
8. Active infection or other medical condition that would make prednisone/prednisolone use contraindicated.
9. Any chronic medical condition requiring a systemic dose of corticosteroid >10 milligrams (mg) prednisone/prednisolone per day.
10. Patients who are considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection.
11. Persistent toxicities (Common Terminology Criteria for Adverse Events [CTCAEs] grade >2) caused by previous cancer therapy, excluding alopecia.
12. Patients with brain metastases. A scan to confirm the absence of brain metastases is not required.
13. Patients with spinal cord compression are excluded unless they are considered to have received definitive treatment for this and have evidence of clinically stable disease for 4 weeks.
14. Patients who are unevaluable for both bone and soft tissue progression
15. Patients who are unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
16. Immunocompromised patients
17. Patients with known active hepatitis infection (ie, hepatitis B or C).
18. Any previous treatment with Polyadenosine 5'diphosphoribose [poly (ADP ribose)] polymerase (PARP) inhibitor, including olaparib.
19. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment. Patients who receive palliative radiotherapy need to stop radiotherapy 1 week before randomisation.
20. Any previous exposure to a Cytochrome P450 (CYP) 17 (17α-hydroxylase/C17,20-lyase) inhibitor (eg, abiraterone, orteronel).
21. Concomitant use of known strong Cytochrome P450 (CYP) 3A inhibitors (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg, ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks.
22. Concomitant use of known strong Cytochrome P450 (CYP) 3A inducers (eg, phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine or St John's wort) or moderate Cytochrome P450 (CYP) 3A inducers (eg, bosentan, efavirenz or modafinil). The required period prior to starting study treatment is 5 weeks for phenobarbital and enzalutamide and 3 weeks for other agents.
23. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
24. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
25. Participation in another clinical study with an investigational product or investigational medical devices within 1 month of randomisation.
26. History of hypersensitivity to olaparib or abiraterone, any of the excipients of olaparib or abiraterone, or drugs with a similar chemical structure or class to olaparib or abiraterone.
27. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca and Merck staff and/or staff at the study site).
28. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
29. Previous randomisation in the present study.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 895 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2026-04-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Saad, MD, Principal Investigator — University of Montreal Hospital Center; Noel Clarke, M.D., Principal Investigator — Christie Hospital Foundation Trust
Locations (117):
- United States (26):
  - Research Site, Birmingham, Alabama
  - Research Site, Anchorage, Alaska
  - Research Site, Tucson, Arizona
  - Research Site, Clovis, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Denver, Colorado
  - Research Site, Lisle, Illinois
  - Research Site, Jeffersonville, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Bozeman, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Paramus, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Rochester, New York
  - Research Site, Syracuse, New York
  - Research Site, Durham, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Myrtle Beach, South Carolina
  - Research Site, Milwaukee, Wisconsin
- Australia (8):
  - Research Site, Box Hill
  - Research Site, Darlinghurst
  - Research Site, Greenslopes
  - Research Site, Herston
  - Research Site, Kingswood
  - Research Site, Kurralta Park
  - Research Site, St Albans
  - Research Site, Waratah
- Research Site, Ghent, Belgium
- Brazil (7):
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Kelowna, British Columbia
  - Research Site, Halifax, Nova Scotia
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Chile (3):
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- France (6):
  - Research Site, Angers
  - Research Site, Besançon
  - Research Site, Caen
  - Research Site, Pierre-Bénite
  - Research Site, Quimper
  - Research Site, Vandœuvre-lès-Nancy
- Germany (10):
  - Research Site, Bergisch Gladbach
  - Research Site, Bremen
  - Research Site, Cologne
  - Research Site, Duisburg
  - Research Site, Freiburg im Breisgau
  - Research Site, Heinsberg
  - Research Site, Mettmann
  - Research Site, Nuremberg
  - Research Site, Nürtingen
  - Research Site, Ulm
- Italy (4):
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Orbassano
  - Research Site, Pavia
- Japan (17):
  - Research Site, Bunkyō City
  - Research Site, Hirakata-shi
  - Research Site, Kanazawa
  - Research Site, Kashihara-shi
  - Research Site, Kawagoe-shi
  - Research Site, Kita-gun
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Miyazaki
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sakura-shi
  - Research Site, Shinjuku-ku
  - Research Site, Toon-shi
  - Research Site, Yokohama
- Netherlands (3):
  - Research Site, Hilversum
  - Research Site, Nijmegen
  - Research Site, Tilburg
- Slovakia (4):
  - Research Site, Bratislava
  - Research Site, Prešov
  - Research Site, Šaľa
  - Research Site, Trenčín
- South Korea (3):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Seoul
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Girona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Karşıyaka
- United Kingdom (5):
  - Research Site, Guildford
  - Research Site, Manchester
  - Research Site, Sheffield
  - Research Site, Southampton
  - Research Site, Swansea

REFERENCES:
- [Derived] Armstrong AJ, Saad F, Oya M, Vianna K, Ozguroglu M, Gedye C, Buchschacher GL Jr, Lee JY, Emmenegger U, Navratil J, Virizuela JA, Salazar A, Maillet D, Uemura H, Hosius C, McGuinness D, Degboe A, Clarke N. Patient-reported Outcomes for Men with Metastatic Castration-resistant Prostate Cancer Who Received Olaparib plus Abiraterone Versus Placebo plus Abiraterone in the Phase 3 PROpel Study. Eur Urol Oncol. 2025 Nov 17:S2588-9311(25)00244-5. doi: 10.1016/j.euo.2025.09.010. Online ahead of print. PMID 41253648
- [Derived] Oya M, Joung JY, Lee JY, Sugimoto M, Choi YD, Hong JH, Uemura H, Nishimura K, Tsumura H, Kawakami S, Hirayama Y, Kwon TG, Kwak C, Suzuki H, Fujita T, Nii M, McGuinness D, Dujka M, Poehlein C, Saad F, Clarke N. Olaparib Plus Abiraterone in Asian Patients With Metastatic Castration-Resistant Prostate Cancer: PROpel Subset Analysis. Cancer Sci. 2025 Jun;116(6):1638-1647. doi: 10.1111/cas.16459. Epub 2025 Mar 18. PMID 40099663
- [Derived] Heiss BL, Chang E, Gao X, Truong T, Brave MH, Bloomquist E, Shah A, Hamed S, Kraft J, Chiu HJ, Ricks TK, Tilley A, Pierce WF, Tang L, Abukhdeir A, Kalavar S, Philip R, Tang S, Pazdur R, Amiri-Kordestani L, Kluetz PG, Suzman DL. US Food and Drug Administration Approval Summary: Talazoparib in Combination With Enzalutamide for Treatment of Patients With Homologous Recombination Repair Gene-Mutated Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2024 May 20;42(15):1851-1860. doi: 10.1200/JCO.23.02182. Epub 2024 Mar 7. PMID 38452327
- [Derived] Clarke NW, Armstrong AJ, Thiery-Vuillemin A, Oya M, Shore N, Loredo E, Procopio G, de Menezes J, Girotto G, Arslan C, Mehra N, Parnis F, Brown E, Schlurmann F, Joung JY, Sugimoto M, Virizuela JA, Emmenegger U, Navratil J, Buchschacher GL, Poehlein C, Harrington EA, Desai C, Kang J, Saad F. Abiraterone and Olaparib for Metastatic Castration-Resistant Prostate Cancer. NEJM Evid. 2022 Sep;1(9):EVIDoa2200043. doi: 10.1056/EVIDoa2200043. Epub 2022 Jun 3. PMID 38319800
- [Derived] Fallah J, Xu J, Weinstock C, Brave MH, Bloomquist E, Fiero MH, Schaefer T, Pathak A, Abukhdeir A, Bhatnagar V, Chiu HJ, Ricks T, John C, Hamed S, Lee C, Pierce WF, Kalavar S, Philip R, Tang S, Amiri-Kordestani L, Pazdur R, Kluetz PG, Suzman D. FDA Approval Summary: Olaparib in Combination With Abiraterone for Treatment of Patients With BRCA-Mutated Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2024 Feb 10;42(5):605-613. doi: 10.1200/JCO.23.01868. Epub 2023 Dec 21. PMID 38127780
- [Derived] Saad F, Clarke NW, Oya M, Shore N, Procopio G, Guedes JD, Arslan C, Mehra N, Parnis F, Brown E, Schlurmann F, Joung JY, Sugimoto M, Sartor O, Liu YZ, Poehlein C, Barker L, Del Rosario PM, Armstrong AJ. Olaparib plus abiraterone versus placebo plus abiraterone in metastatic castration-resistant prostate cancer (PROpel): final prespecified overall survival results of a randomised, double-blind, phase 3 trial. Lancet Oncol. 2023 Oct;24(10):1094-1108. doi: 10.1016/S1470-2045(23)00382-0. Epub 2023 Sep 12. PMID 37714168
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081SC00001&attachmentIdentifier=e550a1c2-29d4-4343-93c6-746de1070fa0&fileName=CSR_Synopsis_redacted_final_pdfa.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081SC00001&attachmentIdentifier=a0849ea5-0997-4872-bbfa-5cfb753f6766&fileName=SAP_redacted_final_all.pdf&versionIdentifier=
- See also: csp_final_compressed — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081SC00001&attachmentIdentifier=2fde9817-51a0-4086-837e-544fa9000666&fileName=CSP_redacted_final_all_(5)-compressed.pdf&versionIdentifier=
- See also: CSR Addendum 1 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081SC00001&attachmentIdentifier=883a40a5-b594-4de5-8dd0-df5f1e7c15aa&fileName=d081sc00001-clinical-study-report-addendum-1.pdf&versionIdentifier=
- See also: CSR addendum 2 - synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D081SC00001&attachmentIdentifier=8900d898-3b43-4dad-bbdd-d636359c02ce&fileName=D081SC00001_CSRaddendum2.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Olaparib 300 mg bd + Abiraterone 1000 mg qd: Patients receive oral treatment with olaparib 300mg twice daily in combination with abiraterone 1000mg once daily
- Placebo bd + Abiraterone 1000 mg qd: Patients receive oral treatment with placebo twice daily in combination with abiraterone 1000mg once daily.
Period: Overall Study
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Started | 399 | 397
Completed | 0 | 0
Not Completed | 399 | 397
Not completed — Death | 168 | 203
Not completed — Other | 2 | 2
Not completed — Failure to meet randomisation criteria | 1 | 1
Not completed — Patient decision | 14 | 10
Not completed — Screen failure | 0 | 1
Not completed — Patients ongoing study at data cut off | 210 | 178
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd | Total
Number analyzed (Participants) | 399 | 397 | 796
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (8.5) | 69.8 (7.9) | 69.1 (8.2)
Age, Customized [Number; unit: Participants]
  >=65 | 269 | 300 | 569
  <65 | 130 | 97 | 227
Sex/Gender, Customized [Number; unit: Participants]
  Male | 399 | 397 | 796
Race/Ethnicity, Customized [Number; unit: Participants]
  HISPANIC OR LATINO | 68 | 63 | 131
  NOT HISPANIC OR LATINO | 310 | 305 | 615
  NOT REPORTED | 21 | 29 | 50
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 1
  ASIAN | 66 | 72 | 138
  BLACK OR AFRICAN AMERICAN | 14 | 11 | 25
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 2 | 0 | 2
  NOT REPORTED | 22 | 30 | 52
  UNKNOWN | 12 | 9 | 21
  WHITE | 282 | 275 | 557
Region of Enrollment [Number; unit: Participants]
  USA | 40 | 34 | 74
  Turkey | 39 | 33 | 72
  Slovakia | 5 | 13 | 18
  Netherlands | 16 | 12 | 28
  Korea, Republic Of | 27 | 29 | 56
  Japan | 36 | 41 | 77
  Italy | 22 | 18 | 40
  United Kingdom | 27 | 22 | 49
  France | 14 | 25 | 39
  Spain | 19 | 24 | 43
  Germany | 14 | 11 | 25
  Czech Republic | 18 | 13 | 31
  Chile | 19 | 25 | 44
  Canada | 17 | 16 | 33
  Brazil | 54 | 46 | 100
  Belgium | 4 | 1 | 5
  Australia | 28 | 34 | 62

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Radiological Progression Free Survival (rPFS) Event by Investigator Assessment
Description: An rPFS event is defined as progression determined by Response Evaluation Criteria in Solid Tumours version 1.1 [RECIST 1.1] and/or Prostate Cancer Working Group 3 [PCWG-3] or death (by any cause in the absence of progression), regardless of whether the patient withdraws from randomised therapy or receives another anticancer therapy prior to progression.
  Per RECIST v1.1, progression is defined as the sum of TLs has a 20% and absolute ≥ 5mm increase from nadir, and/or unequivocal progression in any non target lesions, and/or any new lesion identified.
  Per PCWG3, progression on a bone scan is defined as 2 or more new lesions observed from the first visit after baseline compared to baseline, or from all other visits compared to first visit after baseline. A confirmatory scan is required.
Time Frame: Assessed from date of randomisation to data cut off (DCO1): 30Jul2021 (Approx. 2 years 9 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 399 | 397
Participants | 168 | 226
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Superiority; p < 0.0001, Log Rank — A multiple testing procedure is employed across primary (rPFS) and key secondary endpoints (OS) to strongly control overall type 1 error at 2.5% one-sided; Log rank test stratified by Metastases and Docetaxel at metastatic hormone-sensitive prostate cancer stage using a pre-specified pooling strategy; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.54 to 0.81] — HR and CI calculated using Cox Proportional Hazards model, where a HR < 1 favours olaparib+abiraterone. Stratification factors are the same as those used in the stratified log-rank test

2. Secondary Outcome: Number of Participants With Overall Survival (OS) Event
Description: An OS event is defined as death by any cause, regardless of whether the patient withdraws from randomised therapy or receives another anticancer therapy.
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months). DCO3 is the final data cut-off for the OS analysis and therefore no further updates will be made.
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 399 | 397
Participants | 176 | 205
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Superiority; p = 0.0544, Log Rank — A multiple testing procedure is employed across primary (rPFS) and key secondary endpoints (OS) to strongly control overall type 1 error at 2.5% one-sided. Alpha spend for OS will not exceed 0.02135; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.67 to 1.00] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Time to First Subsequent Anticancer Therapy or Death (TFST) Event
Description: A TFST (excluding radiotherapy) event is defined as the start of the first subsequent anticancer therapy after discontinuation of randomised treatment or death from any cause.
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 399 | 397
Participants | 255 | 285
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Superiority; p = 0.0025, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.64 to 0.90] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Participants With Time to Pain Progression (TTPP) Event
Description: A TTPP event is defined as pain progression based on the Brief Pain Inventory-Short Form (BPI-SF) Item 3 (range 0-10, a higher score indicates worse pain) and opiate analgesic use (Analgesic quantification algorithm [AQA] score, range 0-7, a higher score indicates increased opioid use). For patients who are asymptomatic at baseline (average worst pain score of 0 and not taking opioids): A ≥2 point change from baseline in average (4-7 days) worst pain score observed at 2 consecutive visits or initiation of opioid use; For patients who are symptomatic at baseline (average worst pain score >0 and/or receiving opioids): A ≥2 point change from baseline in average (4-7 days) worst pain score observed at 2 consecutive visits and an average worst pain score ≥4, and no decrease in average opioid use (≥1-point decrease in AQA score from a starting value of ≥2), or increase in opioid use (≥1-point increase, or ≥2-point increase if the starting value is 0) at 2 consecutive follow-up visits.
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 399 | 397
Participants | 68 | 60
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Superiority; p = 0.7456, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.75 to 1.50] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Number of Participants With Opiate Use
Description: An event for opiate use is defined as the first opiate use for cancer related pain.
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Population: Randomised patients who are not on opiates at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 344 | 353
Participants | 58 | 45
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Superiority; p = 0.3099, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.82 to 1.79] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Number of Participants With First Symptomatic Skeletal Related Event (SSRE)
Description: An SSRE event is defined as the first sympomatic skeletal-related event defined by
  * Use of radiation therapy to prevent or relieve skeletal symptoms.
  * Occurrence of new symptomatic pathological bone fractures (vertebral or non-vertebral).
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 399 | 397
Participants | 46 | 51
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Superiority; p = 0.3212, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.55 to 1.22] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Number of Participants With Second Progression or Death (PFS2) Event
Description: An event for PFS2 is defined as the second progression on next-line anticancer therapy or death, whichever occurs earlier.
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 399 | 397
Participants | 103 | 126
Statistical Analysis 1: Comparison: Olaparib 300 mg bd + Abiraterone 1000 mg qd vs Placebo bd + Abiraterone 1000 mg qd; Test type: Superiority; p = 0.0534, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.59 to 0.99] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Brief Pain Inventory-Short Form (BPI-SF)
Description: The BPI-SF is a validated, 15-item domain-specific instrument designed to assess the severity of pain and the impact/interference of pain on daily functions. BPI-SF worst pain, pain severity and pain interference score changes can be a minimum of -10 and a maximum of 10. A negative change from baseline value indicates improvement.
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Population: Full Analysis Set (FAS), only patients with baseline assessment and at least one post treatment assessment are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 330 | 333
Score
  Change from baseline in BPI-SF worst pain | -0.09 (0.093) | 0.03 (0.099)
  Change from baseline in BPI-SF pain severity score | -0.08 (0.071) | -0.02 (0.076)
  Change from baseline in BPI-SF pain interference score | 0.01 (0.074) | 0.13 (0.079)

9. Secondary Outcome: Functional Assessment of Cancer Therapy- Prostate Cancer (FACT-P)
Description: Functional Assessment of Cancer Therapy-Prostate Cancer (FACT-P) total score and Functional Assessment of Cancer Therapy-General (FACT-G) total score.
  Total FACT-P score is the sum of Physical Well-being (PWB), Social Well-being (SWB), Emotional Well-being (EWB), Functional Well-being (FWB) and Prostate cancer subscale (PCS). FACT-P total score change from baseline values can be a minimum of -156 and a maximum of 156. A positive value indicates improvement.
  FACT-G total score is the sum of PWB, SWB, EWB and FWB. FACT-G Total score change from baseline values can be a minimum of -108 and a maximum of 108. A positive value indicates improvement.
Time Frame: Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
Number analyzed (Participants) | 278 | 295
Score
  Change from baseline in FACT-P Total | -5.84 (1.031) | -5.30 (1.060)
  Change from baseline in FACT-G Total | -5.06 (0.766) | -4.35 (0.787)

ADVERSE EVENTS:
Time Frame: Adverse events with an onset date, or worsen, on or after the date of first dose and up to and including 30 days following discontinuation of randomised treatment. Assessed from date of randomisation to data cut off (DCO3): 12Oct2022 (Approx. 3 years 11 months)
Description: Adverse events were assessed based on the Safety population consisting of patients who received treatment (N=794) while all-cause mortality was assessed based on all patients randomized (N=796).
Arm/Group | Olaparib 300 mg bd + Abiraterone 1000 mg qd | Placebo bd + Abiraterone 1000 mg qd
All-Cause Mortality (participants affected / at risk) | 176/399 | 205/397
Serious Adverse Events (participants affected / at risk) | 161/398 | 126/396
Other Adverse Events (participants affected / at risk) | 374/398 | 346/396
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd + Abiraterone 1000 mg qd (N=398) | Placebo bd + Abiraterone 1000 mg qd (N=396)
Acute myocardial infarction (Cardiac disorders) | 4 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 9 (17) | 3 (3)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 5 (5) | 2 (2)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extra-axial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (6) | 4 (5)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 3 (3) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophagia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 23 (29) | 3 (3)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 4 (4)
Loss of consciousness (Nervous system disorders) | 1 (1) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 5 (5) | 2 (2)
Thalamic infarction (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 4 (4)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Prinzmetal angina (Cardiac disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Adventitial cystic disease (Vascular disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Giant cell arteritis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 2 (2)
Limbal stem cell deficiency (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 2 (2)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Asthenia (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 1 (1) | 4 (4)
Fatigue (General disorders) | 3 (3) | 1 (1)
General physical health deterioration (General disorders) | 2 (2) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 2 (2)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholangitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 2 (3)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 1 (1)
Covid-19 (Infections and infestations) | 15 (16) | 10 (10)
Covid-19 pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Cellulitis (Infections and infestations) | 1 (1) | 1 (2)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis b reactivation (Infections and infestations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 2 (2)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia (Infections and infestations) | 11 (13) | 5 (5)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia cryptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 3 (3)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Suspected covid-19 (Infections and infestations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaparib 300 mg bd + Abiraterone 1000 mg qd (N=398) | Placebo bd + Abiraterone 1000 mg qd (N=396)
Upper respiratory tract infection (Infections and infestations) | 21 (22) | 22 (25)
Urinary tract infection (Infections and infestations) | 42 (70) | 33 (41)
Contusion (Injury, poisoning and procedural complications) | 31 (36) | 19 (19)
Fall (Injury, poisoning and procedural complications) | 29 (35) | 28 (35)
Alanine aminotransferase increased (Investigations) | 15 (19) | 27 (30)
Aspartate aminotransferase increased (Investigations) | 16 (18) | 22 (26)
Blood alkaline phosphatase increased (Investigations) | 22 (25) | 21 (24)
Blood creatinine increased (Investigations) | 27 (52) | 19 (26)
Lymphocyte count decreased (Investigations) | 34 (69) | 17 (26)
Weight decreased (Investigations) | 27 (30) | 15 (16)
White blood cell count decreased (Investigations) | 23 (48) | 10 (13)
Decreased appetite (Metabolism and nutrition disorders) | 66 (81) | 31 (33)
Hyperglycaemia (Metabolism and nutrition disorders) | 30 (45) | 27 (36)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 24 (27) | 18 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 33 (54) | 18 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 58 (84) | 77 (116)
Back pain (Musculoskeletal and connective tissue disorders) | 82 (111) | 78 (89)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 34 (44) | 19 (23)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 33 (47) | 28 (31)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (28) | 23 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 38 (46) | 38 (42)
Dizziness (Nervous system disorders) | 49 (53) | 27 (32)
Dysgeusia (Nervous system disorders) | 24 (26) | 7 (7)
Headache (Nervous system disorders) | 39 (44) | 26 (32)
Anaemia (Blood and lymphatic system disorders) | 184 (293) | 67 (93)
Insomnia (Psychiatric disorders) | 31 (35) | 28 (30)
Dysuria (Renal and urinary disorders) | 22 (25) | 18 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (59) | 29 (40)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 (46) | 27 (33)
Hot flush (Vascular disorders) | 35 (37) | 51 (52)
Hypertension (Vascular disorders) | 61 (80) | 74 (97)
Abdominal pain (Gastrointestinal disorders) | 27 (31) | 14 (14)
Abdominal pain upper (Gastrointestinal disorders) | 26 (30) | 16 (18)
Constipation (Gastrointestinal disorders) | 74 (84) | 59 (67)
Diarrhoea (Gastrointestinal disorders) | 80 (109) | 42 (52)
Dyspepsia (Gastrointestinal disorders) | 29 (38) | 17 (20)
Nausea (Gastrointestinal disorders) | 122 (173) | 56 (67)
Lymphopenia (Blood and lymphatic system disorders) | 24 (37) | 10 (11)
Vomiting (Gastrointestinal disorders) | 60 (84) | 36 (42)
Asthenia (General disorders) | 46 (53) | 40 (55)
Fatigue (General disorders) | 112 (131) | 81 (91)
Oedema peripheral (General disorders) | 49 (63) | 50 (62)
Pyrexia (General disorders) | 27 (35) | 19 (24)
Covid-19 (Infections and infestations) | 36 (36) | 25 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03732820/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-14): https://cdn.clinicaltrials.gov/large-docs/20/NCT03732820/SAP_001.pdf